CLINICAL TRIAL: NCT06282731
Title: The Changes of Urine Growth Factors Level in Patients With Benigh Prostate Hyperplasia After Medical Treatment
Brief Title: The Changes of Urine Growth Factors Level
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: En Chu Kong Hospital (Other)
Responsible Party: Principal Investigator, ChungChengWang, Chief of Department of Urology, En Chu Kong Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ECKIRB1020407
Record Dates: First submitted 2019-02-11; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benigh Prostate Hyperplasia(BPH); Urine Growth Factors
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — silodosin; Tamsulosin; Dutasteride; Doxazosin; methanesulfonic acid; Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- urine growth factor (Other): Previous studies have showed that overactive bladder syndrome (urge, frequency, nocturia or urinary incontinence) has been considered as an important factor to predict successful treatment.
  Urine nerve growth factor level, brain-derived neurotrophic factor and endothelium vascular growth factor have been proved as a simple and noninvasive biomarker for diagnosing overactive bladder.
  Interventions: Drug: Silodosin

INTERVENTIONS:
Drug: Silodosin — Indications:Benign prostate hyperplasia
  Other Names: Tamsulosin HCl; Dutasteride; Doxazosin (methanesulfonate); Finasteride

SUMMARY:
The Changes of Urine Growth Factors Level in Patients With Benigh Prostate Hyperplasia after medical treatment.

DETAILED DESCRIPTION:
The prevalence of benign prostate hyperplasia, like medical illness such as hypertension, diabetes mellitus and stroke, increase by age. Benign prostate hyperplasia will cause bothersome lower urinary tract symptoms in the middle and aged male. Previous studies have showed that overactive bladder syndrome (urge, frequency, nocturia or urinary incontinence) has been considered as an important factor to predict successful treatment.

Urine nerve growth factor level, brain-derived neurotrophic factor and endothelium vascular growth factor have been proved as a simple and noninvasive biomarker for diagnosing overactive bladder. As a result, investigator will investigate the changes of these growth factors level in patients with benign prostate hyperplasia before and after three and six-months medical treatment. In addition, investigator can understand whether overactive bladder will have effects on successful medical treatment in patients with benign prostate hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* men with age 50~80 years old
* IPSS>12
* maximal flowrate 5~15ml/sec
* prostate size>20ml
* urine amount>150ml
* patient/family can sigh the inform concent

Exclusion Criteria:

* prostate cancer or suspected prostate cancer(PSA>4ng/ml)
* history of prostate surgery
* free of active urinary tract infection in past 6 months
* patient with any other serious disease considered by investigator not in the condition to enter trials

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-05-31 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Urine growth factors level | One month after medical treatment
  Check Urine growth factors level after one month

SECONDARY OUTCOMES:
Urine growth factors level | Three months after medical treatment
  Check Urine growth factors level afterthree month

OTHER OUTCOMES:
Urine growth factors level | Six months after medical treatment
  Check Urine growth factors level after si xmonth

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Cheng Wang, M.D Ph.D, Principal Investigator — Department of urology,En Chu Nong Hospital
Locations (1):
- En Chu Kong Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams P, Kelleher CJ, Kerr LA, Rogers RG. Overactive bladder significantly affects quality of life. Am J Manag Care. 2000 Jul;6(11 Suppl):S580-90. PMID 11183901
- [Background] De Wachter S, Wyndaele JJ. Frequency-volume charts: a tool to evaluate bladder sensation. Neurourol Urodyn. 2003;22(7):638-42. doi: 10.1002/nau.10160. PMID 14595606
- [Background] Nixon A, Colman S, Sabounjian L, Sandage B, Schwiderski UE, Staskin DR, Zinner N. A validated patient reported measure of urinary urgency severity in overactive bladder for use in clinical trials. J Urol. 2005 Aug;174(2):604-7. doi: 10.1097/01.ju.0000165461.38088.7b. PMID 16006914
- [Background] Romanzi LJ, Groutz A, Heritz DM, Blaivas JG. Involuntary detrusor contractions: correlation of urodynamic data to clinical categories. Neurourol Urodyn. 2001;20(3):249-57. doi: 10.1002/nau.1002. PMID 11385691
- [Background] Apostolidis A, Dasgupta P, Fowler CJ. Proposed mechanism for the efficacy of injected botulinum toxin in the treatment of human detrusor overactivity. Eur Urol. 2006 Apr;49(4):644-50. doi: 10.1016/j.eururo.2005.12.010. Epub 2006 Jan 4. PMID 16426734
- [Background] Hashim H, Abrams P. Is the bladder a reliable witness for predicting detrusor overactivity? J Urol. 2006 Jan;175(1):191-4; discussion 194-5. doi: 10.1016/S0022-5347(05)00067-4. PMID 16406907
- [Background] Vizzard MA. Changes in urinary bladder neurotrophic factor mRNA and NGF protein following urinary bladder dysfunction. Exp Neurol. 2000 Jan;161(1):273-84. doi: 10.1006/exnr.1999.7254. PMID 10683293
- [Background] Yoshimura N. Bladder afferent pathway and spinal cord injury: possible mechanisms inducing hyperreflexia of the urinary bladder. Prog Neurobiol. 1999 Apr;57(6):583-606. doi: 10.1016/s0301-0082(98)00070-7. PMID 10221783
- [Background] Vizzard MA. Neurochemical plasticity and the role of neurotrophic factors in bladder reflex pathways after spinal cord injury. Prog Brain Res. 2006;152:97-115. doi: 10.1016/S0079-6123(05)52007-7. PMID 16198696
- [Background] Seki S, Sasaki K, Igawa Y, et al. Detrusor overactivity induced by increased levels of nerve growth factor in bladder afferent pathways in rats. Neurourol Urodyn. 2003;22:375-377.
- [Background] Lamb K, Gebhart GF, Bielefeldt K. Increased nerve growth factor expression triggers bladder overactivity. J Pain. 2004 Apr;5(3):150-6. doi: 10.1016/j.jpain.2004.01.001. PMID 15106127
- [Background] Yoshimura N, Bennett NE, Hayashi Y, Ogawa T, Nishizawa O, Chancellor MB, de Groat WC, Seki S. Bladder overactivity and hyperexcitability of bladder afferent neurons after intrathecal delivery of nerve growth factor in rats. J Neurosci. 2006 Oct 18;26(42):10847-55. doi: 10.1523/JNEUROSCI.3023-06.2006. PMID 17050722
- [Background] Zvara P, Vizzard MA. Exogenous overexpression of nerve growth factor in the urinary bladder produces bladder overactivity and altered micturition circuitry in the lumbosacral spinal cord. BMC Physiol. 2007 Aug 28;7:9. doi: 10.1186/1472-6793-7-9. PMID 17725832
- [Background] Seki S, Sasaki K, Fraser MO, Igawa Y, Nishizawa O, Chancellor MB, de Groat WC, Yoshimura N. Immunoneutralization of nerve growth factor in lumbosacral spinal cord reduces bladder hyperreflexia in spinal cord injured rats. J Urol. 2002 Nov;168(5):2269-74. doi: 10.1016/S0022-5347(05)64369-8. PMID 12394773
- [Background] Seki S, Sasaki K, Igawa Y, Nishizawa O, Chancellor MB, De Groat WC, Yoshimura N. Suppression of detrusor-sphincter dyssynergia by immunoneutralization of nerve growth factor in lumbosacral spinal cord in spinal cord injured rats. J Urol. 2004 Jan;171(1):478-82. doi: 10.1097/01.ju.0000088340.26588.74. PMID 14665959
- [Background] Cheng CL, Liu JC, Chang SY, Ma CP, de Groat WC. Effect of capsaicin on the micturition reflex in normal and chronic spinal cord-injured cats. Am J Physiol. 1999 Sep;277(3):R786-94. doi: 10.1152/ajpregu.1999.277.3.R786. PMID 10484496
- [Background] Weaver LC, Marsh DR, Gris D, Brown A, Dekaban GA. Autonomic dysreflexia after spinal cord injury: central mechanisms and strategies for prevention. Prog Brain Res. 2006;152:245-63. doi: 10.1016/S0079-6123(05)52016-8. PMID 16198705
- [Background] Steers WD, Kolbeck S, Creedon D, Tuttle JB. Nerve growth factor in the urinary bladder of the adult regulates neuronal form and function. J Clin Invest. 1991 Nov;88(5):1709-15. doi: 10.1172/JCI115488. PMID 1939656
- [Background] Okragly AJ, Niles AL, Saban R, Schmidt D, Hoffman RL, Warner TF, Moon TD, Uehling DT, Haak-Frendscho M. Elevated tryptase, nerve growth factor, neurotrophin-3 and glial cell line-derived neurotrophic factor levels in the urine of interstitial cystitis and bladder cancer patients. J Urol. 1999 Feb;161(2):438-41; discussion 441-2. PMID 9915421
- [Background] Lowe EM, Anand P, Terenghi G, Williams-Chestnut RE, Sinicropi DV, Osborne JL. Increased nerve growth factor levels in the urinary bladder of women with idiopathic sensory urgency and interstitial cystitis. Br J Urol. 1997 Apr;79(4):572-7. doi: 10.1046/j.1464-410x.1997.00097.x. PMID 9126085
- [Background] Liu HT, Kuo HC. Intravesical botulinum toxin A injections plus hydrodistension can reduce nerve growth factor production and control bladder pain in interstitial cystitis. Urology. 2007 Sep;70(3):463-8. doi: 10.1016/j.urology.2007.04.038. PMID 17905097
- [Background] Tuttle JB, Steers WD, Albo M, Nataluk E. Neural input regulates tissue NGF and growth of the adult rat urinary bladder. J Auton Nerv Syst. 1994 Oct;49(2):147-58. doi: 10.1016/0165-1838(94)90134-1. PMID 7806767
- [Background] Dupont MC, Spitsbergen JM, Kim KB, Tuttle JB, Steers WD. Histological and neurotrophic changes triggered by varying models of bladder inflammation. J Urol. 2001 Sep;166(3):1111-8. PMID 11490308
- [Background] Birder LA, Wolf-Johnston A, Griffiths D, Resnick NM. Role of urothelial nerve growth factor in human bladder function. Neurourol Urodyn. 2007;26(3):405-9. doi: 10.1002/nau.20372. PMID 17266135
- [Background] Lommatzsch M, Braun A, Mannsfeldt A, Botchkarev VA, Botchkareva NV, Paus R, Fischer A, Lewin GR, Renz H. Abundant production of brain-derived neurotrophic factor by adult visceral epithelia. Implications for paracrine and target-derived Neurotrophic functions. Am J Pathol. 1999 Oct;155(4):1183-93. doi: 10.1016/S0002-9440(10)65221-2. PMID 10514401
- [Background] Kim JC, Park EY, Seo SI, Park YH, Hwang TK. Nerve growth factor and prostaglandins in the urine of female patients with overactive bladder. J Urol. 2006 May;175(5):1773-6; discussion 1776. doi: 10.1016/S0022-5347(05)00992-4. PMID 16600756
- [Background] Yokoyama T, Kumon H, Nagai A. Correlation of urinary nerve growth factor level with pathogenesis of overactive bladder. Neurourol Urodyn. 2008;27(5):417-20. doi: 10.1002/nau.20519. PMID 17924444
- [Background] Apostolidis A, Popat R, Yiangou Y, Cockayne D, Ford AP, Davis JB, Dasgupta P, Fowler CJ, Anand P. Decreased sensory receptors P2X3 and TRPV1 in suburothelial nerve fibers following intradetrusor injections of botulinum toxin for human detrusor overactivity. J Urol. 2005 Sep;174(3):977-82; discussion 982-3. doi: 10.1097/01.ju.0000169481.42259.54. PMID 16094018
- [Background] Liu HT, Kuo HC. Urinary nerve growth factor level could be a potential biomarker for diagnosis of overactive bladder. J Urol. 2008 Jun;179(6):2270-4. doi: 10.1016/j.juro.2008.01.146. Epub 2008 Apr 18. PMID 18423678
- [Background] Steers WD, Tuttle JB. Mechanisms of Disease: the role of nerve growth factor in the pathophysiology of bladder disorders. Nat Clin Pract Urol. 2006 Feb;3(2):101-10. doi: 10.1038/ncpuro0408. PMID 16470209
- [Background] Abrams PH. Detrusor instability and bladder outlet obstruction. Neurourol Urodyn. 1985;4:317-324.
- [Background] Hyman MJ, Groutz A, Blaivas JG. Detrusor instability in men: correlation of lower urinary tract symptoms with urodynamic findings. J Urol. 2001 Aug;166(2):550-2; discussion 553. doi: 10.1016/s0022-5347(05)65982-4. PMID 11458066
- [Background] Nitti VW, Kim Y, Combs AJ. Voiding dysfunction following transurethral resection of the prostate: symptoms and urodynamic findings. J Urol. 1997 Feb;157(2):600-3. PMID 8996367
- [Background] Digesu GA, Khullar V, Cardozo L, Salvatore S. Overactive bladder symptoms: do we need urodynamics? Neurourol Urodyn. 2003;22(2):105-8. doi: 10.1002/nau.10099. PMID 12579626
- [Background] Liu HT, Kuo HC. Urinary nerve growth factor levels are increased in patients with bladder outlet obstruction with overactive bladder symptoms and reduced after successful medical treatment. Urology. 2008 Jul;72(1):104-8; discussion 108. doi: 10.1016/j.urology.2008.01.069. Epub 2008 Apr 8. PMID 18400272
- [Background] Reitz A, Stohrer M, Kramer G, Del Popolo G, Chartier-Kastler E, Pannek J, Burgdorfer H, Gocking K, Madersbacher H, Schumacher S, Richter R, von Tobel J, Schurch B. European experience of 200 cases treated with botulinum-A toxin injections into the detrusor muscle for urinary incontinence due to neurogenic detrusor overactivity. Eur Urol. 2004 Apr;45(4):510-5. doi: 10.1016/j.eururo.2003.12.004. PMID 15041117
- [Background] Kuo HC. Clinical effects of suburothelial injection of botulinum A toxin on patients with nonneurogenic detrusor overactivity refractory to anticholinergics. Urology. 2005 Jul;66(1):94-8. doi: 10.1016/j.urology.2005.02.002. PMID 15992869
- [Background] Popat R, Apostolidis A, Kalsi V, Gonzales G, Fowler CJ, Dasgupta P. A comparison between the response of patients with idiopathic detrusor overactivity and neurogenic detrusor overactivity to the first intradetrusor injection of botulinum-A toxin. J Urol. 2005 Sep;174(3):984-9. doi: 10.1097/01.ju.0000169480.43557.31. PMID 16094019
- [Background] Werner M, Schmid DM, Schussler B. Efficacy of botulinum-A toxin in the treatment of detrusor overactivity incontinence: a prospective nonrandomized study. Am J Obstet Gynecol. 2005 May;192(5):1735-40. doi: 10.1016/j.ajog.2004.11.052. PMID 15902187
- [Background] Schmid DM, Sauermann P, Werner M, Schuessler B, Blick N, Muentener M, Strebel RT, Perucchini D, Scheiner D, Schaer G, John H, Reitz A, Hauri D, Schurch B. Experience with 100 cases treated with botulinum-A toxin injections in the detrusor muscle for idiopathic overactive bladder syndrome refractory to anticholinergics. J Urol. 2006 Jul;176(1):177-85. doi: 10.1016/S0022-5347(06)00590-8. PMID 16753396
- [Background] Giannantoni A, Di Stasi SM, Nardicchi V, Zucchi A, Macchioni L, Bini V, Goracci G, Porena M. Botulinum-A toxin injections into the detrusor muscle decrease nerve growth factor bladder tissue levels in patients with neurogenic detrusor overactivity. J Urol. 2006 Jun;175(6):2341-4. doi: 10.1016/S0022-5347(06)00258-8. PMID 16697870
- [Background] Patel AK, Patterson JM, Chapple CR. Botulinum toxin injections for neurogenic and idiopathic detrusor overactivity: A critical analysis of results. Eur Urol. 2006 Oct;50(4):684-709; discussion 709-10. doi: 10.1016/j.eururo.2006.07.022. Epub 2006 Aug 4. PMID 16934391
- [Background] Kuo HC. Urodynamic evidence of effectiveness of botulinum A toxin injection in treatment of detrusor overactivity refractory to anticholinergic agents. Urology. 2004 May;63(5):868-72. doi: 10.1016/j.urology.2003.12.007. PMID 15134967
- [Background] Steers WD. Pathophysiology of overactive bladder and urge urinary incontinence. Rev Urol. 2002;4 Suppl 4(Suppl 4):S7-S18. PMID 16986023
- [Background] Liu HT, Chancellor MB, Kuo HC. Urinary nerve growth factor levels are elevated in patients with detrusor overactivity and decreased in responders to detrusor botulinum toxin-A injection. Eur Urol. 2009 Oct;56(4):700-6. doi: 10.1016/j.eururo.2008.04.037. Epub 2008 Apr 30. PMID 18472208
- [Background] Coyne KS, Zhou Z, Thompson C, Versi E. The impact on health-related quality of life of stress, urge and mixed urinary incontinence. BJU Int. 2003 Nov;92(7):731-5. doi: 10.1046/j.1464-410x.2003.04463.x. PMID 14616456
- [Background] Segal JL, Vassallo B, Kleeman S, Silva WA, Karram MM. Prevalence of persistent and de novo overactive bladder symptoms after the tension-free vaginal tape. Obstet Gynecol. 2004 Dec;104(6):1263-9. doi: 10.1097/01.AOG.0000147596.44421.72. PMID 15572487
- [Background] Doo CK, Hong B, Chung BJ, Kim JY, Jung HC, Lee KS, Choo MS. Five-year outcomes of the tension-free vaginal tape procedure for treatment of female stress urinary incontinence. Eur Urol. 2006 Aug;50(2):333-8. doi: 10.1016/j.eururo.2006.04.007. Epub 2006 May 2. PMID 16713066
- [Background] Duckett JR, Basu M. The predictive value of preoperative pressure-flow studies in the resolution of detrusor overactivity and overactive bladder after tension-free vaginal tape insertion. BJU Int. 2007 Jun;99(6):1439-42. doi: 10.1111/j.1464-410X.2007.06842.x. Epub 2007 Apr 5. PMID 17419703
- [Background] Liu HT, Chancellor MB, Kuo HC. Urinary nerve growth factor level could be a biomarker in the differential diagnosis of mixed urinary incontinence in women. BJU Int. 2008 Nov;102(10):1440-4. doi: 10.1111/j.1464-410X.2008.07757.x. Epub 2008 May 16. PMID 18489524
- [Background] Liu HT, Chancellor MB, Kuo HC. Decrease of urinary nerve growth factor levels after antimuscarinic therapy in patients with overactive bladder. BJU Int. 2009 Jun;103(12):1668-72. doi: 10.1111/j.1464-410X.2009.08380.x. Epub 2009 Feb 11. PMID 19220267